CLINICAL TRIAL: NCT05827848
Title: A Prospective, Multicenter, Randomized Withdrawal Trial to Evaluate the Safety and Efficacy of a Percutaneous Peripheral Nerve Stimulation System in Patients With Peripheral Neuropathic Pain
Brief Title: Evaluate the Safety and Efficacy of a Peripheral Nerve Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-22-007
Record Dates: First submitted 2022-11-30; First posted 2023-04-25 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-01

CONDITIONS: Complications; Prosthesis, Nervous System, Peripheral, Pain
Keywords: Peripheral nerve pain
MeSH Terms: conditions — Neurologic Manifestations; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Turn on the machine for continuous nerve stimulation
  Interventions: Device: Percutaneous peripheral nerve stimulation system
- control group (No Intervention): Turn off the machine

INTERVENTIONS:
Device: Percutaneous peripheral nerve stimulation system — All subjects underwent a 7-day baseline assessment (VAS score for at least 4 days) during the screening/baseline period. Eligible subjects underwent PNS surgery and implanted electrode leads and entered the 7-day test period. During the test period, subjects with an average VAS score improvement of ≥30%(VAS score for at least 4 days) will be randomly assigned to the experimental group (on state) or the control group (off state) in a 1:1 ratio for 7 days observation. All subjects were enrolled in the observation period until 28 days after implantation. Safety assessment was performed at a 14-day follow-up after removal of the device.
  Arms: Treatment group

SUMMARY:
This trial was conducted in a prospective, multicenter, randomized withdrawal design at a designated clinical trial facility. The total sample size for this trial is expected to be 59-62 patients.

One to two subjects were conducted in each study center as a preliminary test. A total of about 3-6 subjects were selected for the pre-test. The pre-test subjects used the test equipment (on state) and were not randomized.

The study was divided into screening/baseline period, treatment period (including test period, random withdrawal period and observation period) and follow-up period.

All subjects underwent a 7-day baseline assessment (VAS score for at least 4 days) during the screening/baseline period. Eligible subjects underwent Peripheral Nerve Stimulation(PNS) surgery and implanted electrode leads and entered the 7-day test period. During the test period, subjects with an average VAS score improvement of ≥30%(VAS score for at least 4 days) will be randomly assigned to the experimental group (on state) or the control group (off state) in a 1:1 ratio for 7 days observation. All subjects were enrolled in the observation period until 28 days after implantation. Safety assessment was performed at a 14-day follow-up after removal of the device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, gender unlimited;
* The investigator judged that there was definite peripheral neuropathic pain (chronic and refractory pain in the trunk and extremities, including chronic pain after sternal surgery; Postherpetic neuralgia), suitable for percutaneous peripheral nerve stimulation system treatment;
* Preoperative assessment by neuropathic Pain Scale (DN4) showed that there were related damages or diseases in the peripheral sensory system;
* Patients with poor efficacy or can not tolerate the side effects of treatment after routine treatment;
* Visual analogue scale (VAS)≥50mm within 24 hours before treatment;
* The subject can understand the study purpose, demonstrate sufficient compliance with the study protocol, and be able and willing to sign the informed consent.

Exclusion Criteria:

* Patients who need to be treated with radiofrequency regulation and intrathecal drug infusion;
* Patients who are known to have had heart implants (pacemakers or defibrillators) or other implanted neurostimulators (spinal cord stimulators or deep brain stimulators, etc.);
* Patients with severe psychological and/or psychiatric illness and/or non-therapeutic drug dependence;
* Patients who are expected to undergo MRI within 30 days after PNS implantation;
* Expected to be discharged within 48 hours or less;
* There is known damage to the target nerve or muscle defect in the pain area;
* Patients with known allergies to skin-to-skin contact materials (tape or adhesive);
* Known allergy to anesthetics such as lidocaine;
* Preoperative complications of severe heart, liver, kidney, respiratory diseases and coagulopathy;
* Pregnant or lactating women, or have a birth plan in the next 3 months;
* Is participating in any other drug or medical device clinical trial, or may participate in any other drug or medical device clinical trial after enrollment in this clinical trial;
* The investigator determined that there were other conditions that were not suitable to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference of the mean VAS scores of the experimental group and the control group during the random withdrawal period | 7 days after the wire implantation test period
  (VASEGbase -- VASEGwd) Average - (VASCGbase -- VASCGwd) Average
  Explanation:
  VASEGbase was the mean VAS score of subjects in the experimental group at 4 days before the random withdrawal period.
  VASEGwd was the maximum VAS score of subjects in the experimental group during the random withdrawal period.
  VASCGbase was the mean VAS score of subjects in the control group at 4 days before the random withdrawal period.
  The maximum VAS score of subjects in the VASCGwd control group during the random withdrawal period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ke Ma, PhD, Shanghai, Shanghai Municipality, China